CLINICAL TRIAL: NCT03742362
Title: MRI Study of the Distal Radius Bone Marrow Fat Fraction in Osteoporotic and Healthy Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Uri Nevo (Other)
Collaborators: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Sponsor-Investigator, Uri Nevo, Head of the Bio-Engineering Department, Tel Aviv University
Organization: Tel Aviv University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 0090-18-TLV
Record Dates: First submitted 2018-11-11; First posted 2018-11-15 (Actual); Last update posted 2020-03-03 (Actual); Status verified 2020-03

CONDITIONS: Osteoporosis, Postmenopausal
Keywords: Osteoporosis; MRI; distal radius; postmenopausal
MeSH Terms: conditions — Osteoporosis, Postmenopausal; Osteoporosis

STUDY DESIGN:
Intervention Model Description: 3 groups of women: Group 1: Healthy young women Group 2: Postmenopausal women without Osteoporosis Group 3: Postmenopausal women with Osteoporosis All will undergo the same MRI scans
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Bone marrow fat fraction by MRI (Experimental): MRI scans of distal radius will be performed to all participants to monitor the fat fraction in bone marrow
  Interventions: Device: MRI scans of distal radius

INTERVENTIONS:
Device: MRI scans of distal radius — MRI scans to monitor the fat fraction in the bone marrow of the distal radius

SUMMARY:
The aim of the study is to test whether the distal radius bone marrow show significant difference in the fat fraction in young women compared to post menopausal women with and without osteoporosis.

DETAILED DESCRIPTION:
Patients of the Department of Endocrinology, who routinely perform bone density tests, DXA (Dual Energy X-ray absorpiometry) test on the lumbar spine, proximal femoral and distal radius, will be invited for a visit, and after signing the informed consent form, the following data will be collected: age, BMI, first menstrual period and last menstrual period, family history of osteoporosis, history of osteoporotic fractures, smoking, alcohol use and exercise habits. In addition, blood tests will be performed: calcium phosphate, albumin, alkaline phosphatase, vitamin D level, thyroid function, LH (Luteinizing Hormone) FSH (Follicle Stimulating Hormone), Estradiol, and serum bone turnover index (CTX P1NP). Amount of blood taken: 12 ml The patients will then be sent to the Alfredo Federico Strauss Center for Computerized Neuroimaging at Tel Aviv University for an MRI study of the distal radius. The study results will be analyzed by an expert bone radiologist from the Sourasky Medical Center to reject any kind of pathology (such as a fracture, inflammation, tumor), and further analyzed for bone marrow fat fraction by Tel Aviv University researchers. In the case of abnormal findings, they will be mentioned in the report and the participants will receive recommendations from the appropriate expert.

ELIGIBILITY:
Inclusion Criteria: Women over the age of 45 with regular menstruation should be included in group 1, women over the age of 55 without menstruation for at least one year should be included in groups 2 or 3 according to the results of the bone density test. If T-Score> -2.5 will be included in group 2 and if T-Score <-2.5 they will be included in group 3.

-

Exclusion Criteria: Women with metabolic bone disease, thyroid or pre-thyroid disease, diabetes, chronic steroid use, use of osteoporosis drugs, hormonal therapy, BMI below 20 or over 27, pregnant women and tattooed women in the area under study will not be included in the study.

-

Ages: 45 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Female
Enrollment: 26 (Actual)
Dates: Start 2019-02-02 (Actual); Primary Completion 2019-08-30 (Actual); Study Completion 2019-12-30 (Actual)

PRIMARY OUTCOMES:
Fat fraction in bone marrow | 30 min- 1 hour
  The bone marrow will be studied to determine the percentage of fat

CONTACTS AND LOCATIONS:
Overall Officials: Naftali Stern, Prof, Principal Investigator — Sourasky Medical Center; Uri Nevo, Prof, Principal Investigator — Tel Aviv University; Itzhak Binderman, Prof, Principal Investigator — Tel Aviv University; Yael Schiffenbauer, PhD, Study Director — Tel Aviv University; Vanessa Rouach, MD, Study Director — Sourasky Medical Center; Ido Drukman, MD, Study Director — Sourasky Medical Center
Locations (1):
- Yael Schiffenbauer, Tel Aviv, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] De-Levie TK, Schiffenbauer YS, Druckmann I, Rouach V, Stern N, Binderman I, Nevo U. Quantitative MR Analysis of Changes in the Radius Bone Marrow in Osteoporosis. J Osteoporos. 2023 Dec 27;2023:7861495. doi: 10.1155/2023/7861495. eCollection 2023. PMID 38179189